CLINICAL TRIAL: NCT00484211
Title: NGR008: A Phase II Study of NGR-hTNF Administered as Single Agent Every 3 Weeks or Weekly in Patients Affected by Advanced or Metastatic Hepatocellular Carcinoma (HCC) Previously Treated With no More Than One Systemic Therapeutic Regimen
Brief Title: Study of NGR-hTNF as Single Agent in Patients Affected by Advanced or Metastatic Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AGC Biologics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGR008; 2006-005696-18 (EudraCT Number)
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: NGR-hTNF, Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tumor necrosis factor-alpha, CNGRC fusion protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: NGR-hTNF

INTERVENTIONS:
Drug: NGR-hTNF — iv q3W or q1W 0.8 mcg/sqm NGR-hTNF

SUMMARY:
The main objective of the trial is to document the progression free survival (PFS) in advanced or metastatic hepatocellular carcinoma patients treated with NGR-hTNF as single agent.

Safety will be established by clinical and laboratory assessment according to NCI-CTC criteria

DETAILED DESCRIPTION:
This is a phase II, open-label, non-randomized study that will be conducted in patients affected by advanced or metastatic Hepatocellular Carcinoma (HCC) previously treated with no more than one systemic therapeutic regimen, that will be conducted using Simon's two-stage design method.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years affected by advanced or metastatic HCC previously treated with no more than one systemic therapeutic regimen
* Histologically confirmed HCC not amenable to curative surgery
* Child-Pugh scale class A
* ECOG Performance status 0 - 1
* Patients in progression disease at study entry CT documented
* Adequate baseline bone marrow, hepatic and renal function, defined as follows:

  * Neutrophils > 1.5 x 10^9/L and platelets > 100 x 10^9/L
  * Bilirubin < 2 x ULN
  * Transaminases < 3 x ULN
* Absence of any conditions in which hypervolaemia and its consequences (e.g. increased stroke volume, elevated blood pressure) or haemodilution could represent a risk for the patient (reference appendix "Technical data sheet human albumin")
* Normal cardiac function and absence of uncontrolled hypertension
* Patients must give written informed consent

Exclusion criteria:

* Decompensated cirrhosis (Child-Pugh score >7)
* Concurrent anticancer therapy
* Patients may not receive any other investigational agents while on study
* Clinical signs of CNS involvement
* Patients with active or uncontrolled systemic disease/infections or with serious illness or medical conditions, which is incompatible with the protocol
* Known hypersensitivity/allergic reaction to human albumin preparations or to any of the excipients
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol
* Pregnancy or lactation. Patients - both males and females - with reproductive potential (i.e. menopausal for less than 1-year and not surgically sterilized) must practice effective contraceptive measures throughout the study. Women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-12; Primary Completion 2011-11 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Antitumour activity defined as progression free survival (PFS) | during the study

SECONDARY OUTCOMES:
Tumor growth control rate (TGCR) according to WHO criteria | during the study
Pharmacokinetics in patients treated with weekly schedule | during treatment
Safety | during the study
Overall survival (OS) | During the treatment and during the follow-up
Experimental imaging study (DCE-MRI) | During the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Lambiase, MD, Study Director — AGC Biologics S.p.A.
Locations (3):
- Italy (3):
  - Fondazione San Raffaele del Monte Tabor, Milan, Milan
  - Istituto Europeo Oncologico, Milan, Milan
  - Istituto Clinico Humanitas, Rozzano, Milan

REFERENCES:
- [Result] Santoro A, Pressiani T, Citterio G, Rossoni G, Donadoni G, Pozzi F, Rimassa L, Personeni N, Bozzarelli S, Rossoni G, Colombi S, De Braud FG, Caligaris-Cappio F, Lambiase A, Bordignon C. Activity and safety of NGR-hTNF, a selective vascular-targeting agent, in previously treated patients with advanced hepatocellular carcinoma. Br J Cancer. 2010 Sep 7;103(6):837-44. doi: 10.1038/sj.bjc.6605858. Epub 2010 Aug 17. PMID 20717115